CLINICAL TRIAL: NCT04093089
Title: Clinical Study Of The Bionode System In Subjects With Elevated Intraocular Pressure (IOP)
Brief Title: Clinical Study Of The Bionode System In Subjects With Elevated IOP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bionode, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00029387
Record Dates: First submitted 2019-08-27; First posted 2019-09-17 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Unmedicated IOP Before and After Treatment

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental)
  Interventions: Device: Bionode IOP Lowering System
- Control Group (Placebo Comparator)
  Interventions: Device: Bionode IOP Lowering System

INTERVENTIONS:
Device: Bionode IOP Lowering System — Patients wearing Bionode spectacles and customized contact lens and will receive stimulation at 50 Hz, 100 µs, up to 150 µA for 2 hours.
  Arms: Test Group
Device: Bionode IOP Lowering System — Control: No stimulation
  Arms: Control Group

SUMMARY:
The primary objective of this study is to evaluate the safety and effectiveness of the Bionode IOP lowering system in eyes with elevated IOP. The contact lens being studied is similar to an ordinary contact lens that is worn to correct nearsightedness. But the study contact lens has been designed with a thin gold coil around the outside edge of the lens. This design helps deliver a low amount of energy to the eye, which is expected to help lower the pressure inside of the eye. The study contact lens is activated by a pair of glasses (Bionode spectacles) that you wear to apply the treatment to your eye. The study contact lens is only activated when the study glasses are activated.

DETAILED DESCRIPTION:
Subjects will be randomized in 1:1 ratio into two groups, designated Group A and Group B. During the study, randomized subjects will be fitted with a pair of study contact lenses, only one of which is embedded with a gold coil to receive electrical stimulation from the study spectacles, in the study eye. Subjects will also wear optical spectacles (study spectacles) that deliver the electrical stimulus the study contact lenses.

Group A will receive electrical stimulation (test group), and Group B will not receive electrical stimulation (control group). Baseline IOP will be recorded prior to the 2-hours stimulation, and will be repeated post-therapy, at increments of 5 minutes, 30 minutes, 60 minutes, and 2 hours from the conclusion of stimulation. The total duration of participation for each subject is up to approximately 5 weeks. The total expected duration of the clinical trial is approximately 4 months.

ELIGIBILITY:
Inclusion Criteria:

1. Subject ability and willingness to read, comprehend and signed the informed consent form.
2. Subject willingness to comply with study instructions, agreement to make all office appointments, and complete the entire course of the study.
3. Clinical diagnosis of primary open-angle glaucoma (POAG) or ocular hypertension (OHT) with IOP > 22 mmHg.
4. Subjects > 22 years of age at the time of the screening examination.
5. Central corneal thickness of > 450 µm and < 650 µm in study eye
6. Best-corrected visual acuity (BCVA) or pinhole visual acuity (Snellen) of 20/100 or better in study eye.
7. Subjects with an angle of grade 2 or above via the Shaffer grading system

Exclusion Criteria:

1. Angle-closure glaucoma, neovascular glaucoma, traumatic glaucoma or iridocorneal endothelium syndrome in either eye
2. Corneal endothelial dysfunction or abnormalities (e.g., Fuchs' Corneal Dystrophy) in either eye
3. Known sensitivity to any products (e.g., contact lens) required for the study procedures
4. A vertical cup to disc ratio of > 0.8, or notched optic nerve head rim in either eye
5. Visual defect within 10 degrees of fixation or mean deviation of worse than -10 dB
6. History of complications, trauma or disease in the nasolacrimal area.
7. Structural lid abnormalities (i.e., ectropion, entropion) in study eye
8. Active lid disease in either eye (i.e., moderate or severe blepharitis, Meibomian gland dysfunction) that requires medical treatment
9. History of chronic/recurrent inflammatory eye disease (i.e., scleritis, uveitis, herpes keratitis) in either eye
10. Any ophthalmic surgical procedures (i.e., glaucoma laser, minimally invasive glaucoma surgery, refractive, etc.) in study eye within the last six months or will require ophthalmic surgery before completing study
11. History of penetrating keratoplasty in study eye
12. Use of a contact lens in either eye at any time during the study period
13. Uncontrolled diabetic retinopathy, branch retinal vein occlusion or central retinal vein occlusion in either eye
14. Any systemic medication [i.e., beta-blocker, carbonic anhydrase inhibitors, corticosteroids (including dermal), etc.], that may have an effect on the subject's IOP, or who will require its use during the study period (Note: an inhaled steroid, systemic beta-blocker or β-adrenoceptor antagonist may be permitted, providing the subject has maintained a stable dosage regimen for at least the last three months)
15. Women who are pregnant or lactating.
16. Severe dry eyes.
17. LASIK surgery.
18. Subject currently participating or has participated within the last 30 days prior to the start of this study in a drug, device or other investigational research study
19. Subject who cannot be successfully fitted with Bionode spectacles and wear contact lenses (if applicable) at the Baseline Visit (day 0)

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-07-17 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure (mmHg) | 0 min (baseline), 5 min, 30 min, 60 min, and 120 min post treatment
  The primary effectiveness outcome is defined unmedicated IOP after treatment, at 0 min (baseline), 5 min, 30 min, 60 min, and 120 min. An area under the curve will be calculated from the IOP measures at the 5 time points.
Number of patients with treatment related adverse events | 1 month post treatment
  Incidence of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Ayda Shahidi, PhD, Study Director — Prism Eye Institute
Locations (1):
- Prism Eye Institue, Oakville, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided